CLINICAL TRIAL: NCT00929201
Title: An Open-Label, Randomized, Two-Period Crossover Definitive Bioequivalence Study With the Final Marketed Image (FMI) Sitagliptin/Metformin Fixed-Dose Combination (FDC) Tablet and Co-Administration of the Sitagliptin and Metformin Individual Tablets After Consumption of a High-Fat Meal in Healthy Adult Subjects
Brief Title: Sitagliptin/Metformin Fed Bioequivalence Study (0431A-080)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0431A-080; MK-0431A-080 (Other: Merck protocol number); 2009_607 (Other: Merck registration number)
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2010-02-01 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sita + Met then Sita/Met FDC (Active Comparator): Participants receive sitagliptin (Sita) 50 mg and metformin (Met) 500 mg individual tablets administered concomitantly as a single dose during Period 1 followed by a 7-day washout followed by sitagliptin/metformin (Sita/Met) 50/500 mg FDC tablet administered as a single dose during Period 2.
  Interventions: Drug: Sitagliptin phosphate/metformin hydrochloride FDC; Drug: Sitagliptin phosphate; Drug: Metformin hydrochloride
- Sita/Met FDC then Sita + Met (Active Comparator): Participants receive sitagliptin/Metformin 50 mg/500 mg FDC tablet administered as a single dose during Period 1 followed by a 7-day washout followed by sitagliptin 50 mg and metformin 500 mg individual tablets administered concomitantly as a single dose during Period 2.
  Interventions: Drug: Sitagliptin phosphate/metformin hydrochloride FDC; Drug: Sitagliptin phosphate; Drug: Metformin hydrochloride

INTERVENTIONS:
Drug: Sitagliptin phosphate/metformin hydrochloride FDC — Single dose sitagliptin/metformin 50/500 mg FDC tablet after consumption of a high-fat meal in one of two treatment periods.
Drug: Sitagliptin phosphate — Single dose sitagliptin 50 mg tablet after consumption of a high-fat meal in one of two treatment periods.
Drug: Metformin hydrochloride — Single dose metformin 500 mg tablet after consumption of a high-fat meal in one of two treatment periods.

SUMMARY:
This study will demonstrate the bioequivalence of metformin after single dose administration of sitagliptin/metformin 50/500 mg fixed dose combination (FDC) tablet and concomitant administration of single doses of sitagliptin 50 mg and metformin 500 mg as individual tablets after consumption of a high-fat meal.

ELIGIBILITY:
Inclusion Criteria:

* is in good health
* is a nonsmoker
* is willing to follow all study guidelines

Exclusion Criteria:

* has or has a history of any illness or condition that might confound the results of the study or make participation unsafe for the participant
* is a nursing mother
* is unwilling to consume the required high-fat breakfast

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Sita + Met Then Sita/Met FDC: Sitagliptin 50 mg and metformin 500 mg individual tablets administered concomitantly as a single dose during Period 1 followed by a 7-day washout followed by sitagliptin/metformin (Sita/Met) 50/500 mg fixed-dose combination (FDC) tablet administered as a single dose during Period 2.
- Sita/Met FDC Then Sita + Met: Sitagliptin/Metformin 50 mg/500 mg FDC tablet administered as a single dose during Period 1 followed by a 7-day washout followed by sitagliptin 50 mg and metformin 500 mg individual tablets administered concomitantly as a single dose during Period 2.
Period: Period 1
Arm/Group | Sita + Met Then Sita/Met FDC | Sita/Met FDC Then Sita + Met
Started | 30 | 31
Completed | 30 | 30
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: 7-day Washout
Arm/Group | Sita + Met Then Sita/Met FDC | Sita/Met FDC Then Sita + Met
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sita + Met Then Sita/Met FDC | Sita/Met FDC Then Sita + Met
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All randomized participants
Arm/Group | All Participants
Number analyzed (Participants) | 61
Age, Continuous [Mean (Full Range); unit: Years] | 32.4 [18 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 29
Height [Mean (Full Range); unit: Centimeters] | 164.9 [150.0 to 184.0]
Weight [Mean (Full Range); unit: Kilograms] | 73.0 [45.9 to 102.3]

OUTCOME MEASURES:

1. Primary Outcome: Plasma Area Under the Curve (AUC(0 to Infinity)) for Metformin
Description: Serum samples were used to determine the AUC from time 0 to infinity for metformin.
Time Frame: Predose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 32, 48, and 72 hours postdose
Population: All participants who completed and who had pharmacokinetic data available from at least one treatment period
Measure: Least Squares Mean (Standard Deviation); unit: μg * hr/mL
Groups:
- Sita + Met: Sitagliptin 50 mg and metformin 500 mg individual tablets administered concomitantly as a single dose
- Sita/Met FDC: Sitagliptin/Metformin 50 mg/500 mg final marketed image (FMI) FDC tablet administered as a single dose
Arm/Group | Sita + Met | Sita/Met FDC
Number analyzed (Participants) | 60 | 60
μg * hr/mL | 7.65 (1.39) | 7.45 (1.48)
Statistical Analysis 1: Comparison: Sita + Met vs Sita/Met FDC; Least-Squares Mean Ratio calculated as Sitagliptin/Metformin 50/500 mg FDC tablet divided by Sitagliptin 50 mg and metformin 500 mg individual tablets; Test type: Non-Inferiority or Equivalence — The FMI sitagliptin/metformin 50/500 mg FDC tablet and coadministration of corresponding doses of sitagliptin and metformin as individual tablets after consumption of a standard high-fat breakfast will be bioequivalent for metformin based on assessment of the AUC0-∞ for metformin [i.e., the true metformin AUC0-∞GMR (sitagliptin/metformin 50/500 mg FDC tablet/co-administration of sitagliptin and metformin as individual tablets will be contained within (0.80, 1.25)]; Least-Squares Mean Ratio = 0.97, 90% CI [0.95 to 1.00]

2. Secondary Outcome: Peak Plasma Concentration (Cmax) of Metformin
Description: Serum samples were used to determine the maximum concentration for metformin.
Time Frame: Predose and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 16, 24, 32, 48, and 72 hours postdose
Population: All participants who completed and who had pharmacokinetic data available from at least one treatment period
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Groups:
- Sita/Met FDC: Sitagliptin/Metformin 50 mg/500 mg FMI FDC tablet administered as a single dose
Arm/Group | Sita + Met | Sita/Met FDC
Number analyzed (Participants) | 60 | 60
ng/mL | 929 (181) | 887 (187)
Statistical Analysis 1: Comparison: Sita + Met vs Sita/Met FDC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — The FMI sitagliptin/metformin 50/500 mg FDC tablet and co-administration of corresponding doses of sitagliptin and metformin as individual tablets after consumption of a standard high-fat breakfast will be bioequivalent for metformin based on assessment of the Cmax for metformin [i.e., the true metformin Cmax GMR (sitagliptin/metformin 50/500 mg FDC tablet/ co-administration of sitagliptin and metformin as individual tablets will be contained within (0.80, 1.25)]; Least-Squares Mean Ratio = 0.95, 90% CI [0.93 to 0.98]

ADVERSE EVENTS:
Time Frame: Up to 24 days (including 14 days after administration of study drug in the last treatment period)
Description: All participants as treated defined as all participants who received at least one dose of study drug
Arm/Group | Sita + Met | Sita/Met FDC
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/61
Other Adverse Events (participants affected / at risk) | 2/60 | 6/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sita + Met (N=60) | Sita/Met FDC (N=61)
Headache (Nervous system disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.